CLINICAL TRIAL: NCT02580006
Title: A Randomized, Double-blind, Active Control, Single Dosing, Crossover Clinical Trial to Investigate the Pharmacokinetics of EPORON® and EPREX® After Subcutaneous Administration in Healthy Male Volunteers
Brief Title: To Investigate the Pharmacokinetics of EPORON® and EPREX® After Subcutaneous Administration in Healthy Male Volunteers
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Dong-A ST Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: DA3285_SC_I
Record Dates: First submitted 2015-10-13; First posted 2015-10-20 (Estimated); Last update posted 2015-10-20 (Estimated); Status verified 2015-10

CONDITIONS: Healthy
MeSH Terms: interventions — Epoetin Alfa

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- EPORON→EPREX (Experimental): EPORON PFS(PreFilled Syringe) 4000 IU/0.4 mL(Erythropoietin alfa 4000 IU) will be administered subcutaneously after 10 hours fasting on Day 1.
  And wash out for 4 weeks. EPREX INJ.(Injection) 4000 IU(Erythropoietin alfa 4000 IU) will be administered subcutaneously after 10 hours fasting on Day 29.
  Interventions: Drug: EPORON; Drug: EPREX
- EPREX→EPORON (Experimental): EPREX INJ. 4000 IU(Erythropoietin alfa 4000 IU) will be administered subcutaneously after 10 hours fasting on Day 1.
  And wash out for 4 weeks. EPORON PFS 4000 IU/0.4 mL(Erythropoietin alfa 4000 IU) will be administered subcutaneously after 10 hours fasting on Day 29.
  Interventions: Drug: EPORON; Drug: EPREX

INTERVENTIONS:
Drug: EPORON — single dose administration subcutaneously
  Other Names: EPORON PFS 4000 IU/0.4 mL (Erythropoietin alfa 4000 IU)
Drug: EPREX — single dose administration subcutaneously
  Other Names: EPREX INJ. 4000 IU (Erythropoietin alfa 4000 IU)

SUMMARY:
This Phase I study is to compare pharmacokinetics, safety and pharmacodynamics of EPORON and EPREX after single subcutaneous administration.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteers between the ages of 19~50 at the time of screening
* Weight between 55.0kg~90.0kg with BMI of 18.0~27.0
* Voluntarily participants who agree to observe the precautions in writing after receiving a complete explanation of this trial

Exclusion Criteria:

* History of clinically significant illness related to liver (including viral hepatitis), kidney, nervous system, immune system, respiratory system, endocrine system, cardiovascular system, blood system and tumor as well as mental illness (mood disorder, obsessive-compulsive disorder, etc.)
* Hypersensitivity or clinically significant hypersensitivity to the drug (e.g. aspirin, antibiotics, etc.)
* Those whose results meet more than one of the followings in the screening including re-test; Hemoglobin level below 12g/dL or over 17g/dL, Vitamin B12 level below 200pg/mL, Ferritin level below 21.8ng/mL, Transferrin level below 190mg/dL, Reticulocyte, erythrocytes, platelets or serum potassium level over normal range
* Positive on the HIV antibody, HBsAg, HCV(Hepatitis C Virus) antibody tests
* Those whose vital signs measured in sitting position after resting over 3 minutes meet more than one of the following; Systolic BP below 90mmgHg or over 160mmgHg, Diastolic BP below 50mmgHg or over 100mmgHg, Pulse rate over 100
* History of drug abuse, or tested positive in the urine drug screening
* Administration of EPO(erythropoietin), darbepoetin or other EPO protein supply, immunoglobulin within 3 months from the scheduled first dose
* Hypersensitivity to EPO, darbepoetin or excipient in the test drug or anaphylactic reaction towards iron supplement
* Those who received the following diagnosis within 6 months from the screening; Hemoglobinopathy (e.g., homozygous sickle-cell disease, thalassemia of all kinds), Chronic or uncontrollable inflammatory diseases (e.g., rheumatoid arthritis, systemic erythematosus)
* Those who took any ETC(Ethical) drugs or herbal medicine within 2 weeks, or any OTC(Over-the-counter) drugs or vitamins within a week from the scheduled first dose (However, they may be included as the trial subjects at the discretion of the investigator if other conditions are satisfactory.)
* Those who participated other clinical trials and was administered other drugs within 3 months from the scheduled first dose
* Those who bled over 400mL or donated blood within 8 weeks from the scheduled first dose
* Those who have continued drinking (exceeding 21 units/week, 1 unit = 10g of pure alcohol) or who can't abstain from alcohol during the trial period
* Those who have smoked over 10 cigarettes daily in average for the last 3 months or who can't renounce smoking during the trial period
* Those who have ingested grapefruit or caffeine containing food within 3 days from the scheduled first dose or who can't abstain from the during the trial period.
* Those who are preparing for pregnancy or who do not agree with contraception during the trial period
* Those with peculiar eating habits or who can't have meals provided by the hospital
* Those who are considered inappropriate for the trial by the trial investigator based on the result of clinical laboratory test or due to other reasons

Ages: 19 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Estimated)
Dates: Start 2015-11; Primary Completion 2016-01 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Area Under Curve last(AUClast) of Erythropoietin | Twice every 10 minutes within 1hr before administration (day 1/day 29); immediately before administration; 1, 2, 4, 6, 8, 10, 12, 14, 16, 24, 36, 48, 72, 96, 120 (day 6/day 34), 144 (day 7/day 35) hrs after administration for each period
Maximum of concentration(Cmax) of Erythropoietin | Twice every 10 minutes within 1hr before administration (day 1/day 29); immediately before administration; 1, 2, 4, 6, 8, 10, 12, 14, 16, 24, 36, 48, 72, 96, 120 (day 6/day 34), 144 (day 7/day 35) hrs after administration for each period
Reticulocyte count (%) compared to baseline | Twice every 10 minutes within 1hr before administration (day 1/day 29); immediately before administration; 12, 24, 48, 72, 96, 120 (day 6/day 34), 144 (day 7/day 35), 216 (day 10/day 38), 312 (day 14/day 42) hrs after administration for each period
  The absolute difference from the most increased case and its relative percentage (%) when comparing the results before administration

SECONDARY OUTCOMES:
Time of maximum concentration(Tmax) of Erythropoietin | Twice every 10 minutes within 1hr before administration (day 1/day 29); immediately before administration; 1, 2, 4, 6, 8, 10, 12, 14, 16, 24, 36, 48, 72, 96, 120 (day 6/day 34), 144 (day 7/day 35) hrs after administration for each period
Terminal half-life(t1/2) of Erythropoietin | Twice every 10 minutes within 1hr before administration (day 1/day 29); immediately before administration; 1, 2, 4, 6, 8, 10, 12, 14, 16, 24, 36, 48, 72, 96, 120 (day 6/day 34), 144 (day 7/day 35) hrs after administration for each period
Area Under Curve infinity(AUCinf) of Erythropoietin | Twice every 10 minutes within 1hr before administration (day 1/day 29); immediately before administration; 1, 2, 4, 6, 8, 10, 12, 14, 16, 24, 36, 48, 72, 96, 120 (day 6/day 34), 144 (day 7/day 35) hrs after administration for each period
Apparent Clearance(CL/F) of Erythropoietin | Twice every 10 minutes within 1hr before administration (day 1/day 29); immediately before administration; 1, 2, 4, 6, 8, 10, 12, 14, 16, 24, 36, 48, 72, 96, 120 (day 6/day 34), 144 (day 7/day 35) hrs after administration for each period
Mean Residence Time last(MRTlast) of Erythropoietin | Twice every 10 minutes within 1hr before administration (day 1/day 29); immediately before administration; 1, 2, 4, 6, 8, 10, 12, 14, 16, 24, 36, 48, 72, 96, 120 (day 6/day 34), 144 (day 7/day 35) hrs after administration for each period
Hemoglobin | Twice every 10 minutes within 1hr before administration (day 1/day 29); immediately before administration; 12, 24, 48, 72, 96, 120 (day 6/day 34), 144 (day 7/day 35), 216 (day 10/day 38), 312 (day 14/day 42) hrs after administration for each period
Hematocrit | Twice every 10 minutes within 1hr before administration (day 1/day 29); immediately before administration; 12, 24, 48, 72, 96, 120 (day 6/day 34), 144 (day 7/day 35), 216 (day 10/day 38), 312 (day 14/day 42) hrs after administration for each period
RBC count | Twice every 10 minutes within 1hr before administration (day 1/day 29); immediately before administration; 12, 24, 48, 72, 96, 120 (day 6/day 34), 144 (day 7/day 35), 216 (day 10/day 38), 312 (day 14/day 42) hrs after administration for each period

CONTACTS AND LOCATIONS:
Overall Officials: Kyung-sang Yu, MD, Ph.D, Principal Investigator — Clinical Pharmacology Class of Seoul National University College of Medicine / Clinical Pharmacology of Seoul National University Hospital; In-jin Jang, MD, Ph.D, Study Director — Clinical Pharmacology Class of Seoul National University College of Medicine / Clinical Pharmacology of Seoul National University Hospital; Hyung-gi Lee, MD, Ph.D, Study Director — Clinical Pharmacology Class of Seoul National University College of Medicine / Clinical Pharmacology of Seoul National University Hospital; Ju-yeon Cho, Ph.D, Study Director — Clinical Pharmacology Class of Seoul National University College of Medicine / Clinical Pharmacology of Seoul National University Hospital; Seung-hwan Lee, MD, Ph.D, Study Director — Seoul National University Hospital Clinical Trials Center / Clinical Pharmacology of Seoul National University Hospital
Locations (1):
- Seoul National University Hospital Clinical Trials Center, Seoul, South Korea